CLINICAL TRIAL: NCT01743417
Title: Computerized Cognitive Rehabilitation in Children After Severe Malaria
Acronym: CM_CCRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Michigan State University (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01HD064416-01A1 (NIH)
Record Dates: First submitted 2012-09-05; First posted 2012-12-06 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Malaria
Keywords: Cognitive rehabilitation; malaria; neuropsychology; attention; working memory
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive intervention (Experimental): Children in this arm will receive computerised cognitive rehabilitation training for 24 sessions lasting 45 minutes. The Captain's log brain training software is programmed to increase in difficulty as child progresses through the training levels.
  Interventions: Behavioral: Computerised cognitive rehabilitation training
- Active control (Active Comparator): Children in this arm will receive 24 sessions of computerised cognitive rehabilitation training. Captain's log, the brain training software will not be programmed to increase in difficulty with each successive level in this arm.
  Interventions: Behavioral: Computerised cognitive rehabilitation training
- Passive control (No Intervention): No computer training or games will be provided to this group

INTERVENTIONS:
Behavioral: Computerised cognitive rehabilitation training — 24 sessions of computerised bran training will be provided for 8 weeks (+/-2) with about 3 sessions per week to the intervention arm and active control arms. The program will be programmed to increases in difficulty for the intervention arm. In the active control arms, the difficulty level will not change.
  Other Names: Captain's Log
  Arms: Active control; Cognitive intervention

SUMMARY:
Brain training exercises will be provided to children who survived an episode of severe malaria. These children will be given assessments for cognition, behaviour and executive functions before and after the brain training exercises.

DETAILED DESCRIPTION:
Background:

Our Fogarty "Brain Disorders" R21 study findings demonstrated that attention and working memory deficits persist in one out of four children with cerebral malaria (CM) (Boivin et al., 2007; John, Bangirana et al., 2008). Uganda has one of the highest incidences of malaria worldwide (~480/1000) with about 10% of these incidents becoming severe and over 90% of such cases occurring in children (Snow, Guerra, Noor, Myint, & Hay, 2005). This results in an estimated 80 thousand new cases each year of Ugandan children with mild to severe neurocognitive impairment from this disease. Such impairment will likely compromise their school performance, impede their activities of daily living, and lessen their future economic opportunities.

There is no known treatment intervention during acute illness to prevent CM brain-injury effects (Abubakar et al., 2007). Nor are neurocognitive rehabilitative treatment programs available in low-resource settings for affected children. However, we have successfully piloted a computerized cognitive rehabilitation therapy (CCRT) intervention to specifically improve attention, visual-spatial learning, and psychosocial adjustment (domains shown most affected by CM in our previous studies) with school-age Ugandan CM survivors (Bangirana, Giordani et al., 2009). This evidence justifies an R01 for further study.

The present application proposes a randomized control trial (RCT) to further establish that CCRT can improve attention, working memory, aspects of executive functioning, and psychosocial adjustment in pediatric CM survivors. Such programs are already being used extensively with children with developmental disabilities (e.g., Attention Deficit Hyperactivity Disorder, learning disorders) and brain injury in high-income countries. The evidence from RCT studies for these interventions is strong enough to warrant the evaluation of CCRT for at-risk African children (Bangirana, Idro, John, & Boivin, 2006; Boivin & Giordani, 2009). CCRT could also then be extended to a variety of other infectious diseases causing brain injury and persisting neurocognitive deficits to children in this setting (e.g., HIV, schistosomiasis, meningitis, encephalitis, and neurocysticercosis).

Objectives:

1. To evaluate the effectiveness of CCRT in improving neuropsychological performance and psychiatric outcomes in Ugandan children who survive severe malaria.
2. To evaluate whether severity of malaria illness (e.g., immunological brain inflammation, EEG abnormalities) is predictive of neuropsychological benefit from CCRT.
3. METHODS

Study design:

Randomized controlled trial

Study Population:

Our proposed study groups of children aged 5 to 12 years will consist of 150 children with severe malaria (either cerebral malaria or severe malaria anemia). From the homes of these severe malaria children, we will also recruit 1 sibling (or neighbor child) 5 to 12 years of age without a history of cerebral malaria or other known infectious disease that could cause brain injury (Community Controls from Home: CC children N = 150).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 5 to 12 years of age;
2. Signed consent from the parent/guardian, assent from children aged 7 years and older;
3. Completion of their 24 months testing in the parent study (MUREC no 2008-033).

Exclusion Criteria:

1. CM: elevated cerebrospinal fluid protein, white blood cells or red blood cells
2. Severe malarial anemia: history of coma, impaired consciousness, repeated seizures, other brain disorder, and developmental delay. Additional exclusion criteria for CC group:

   * any active illness; recent illness or recovery from illness;
   * chronic illness requiring medical care; -) medical abnormalities on screening history or physical exam.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-08-23 (Actual); Study Completion 2016-08-23 (Actual)

PRIMARY OUTCOMES:
Executive attention | Measured at 12 months post-intervention
  Executive attention will be measured by the Test of Variables of Attention

SECONDARY OUTCOMES:
Working memory | Measured at 12 months post-intervention
  Working memory will be measured by the Kaufman Assessment Battery for Children second edition

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Boivin, PhD, Principal Investigator — Michigan State University; Noeline Nakasujja, PhD, Principal Investigator — Makerere University
Locations (1):
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bangirana P, Allebeck P, Boivin MJ, John CC, Page C, Ehnvall A, Musisi S. Cognition, behaviour and academic skills after cognitive rehabilitation in Ugandan children surviving severe malaria: a randomised trial. BMC Neurol. 2011 Aug 4;11:96. doi: 10.1186/1471-2377-11-96. PMID 21816079
- [Background] Bangirana P, Giordani B, John CC, Page C, Opoka RO, Boivin MJ. Immediate neuropsychological and behavioral benefits of computerized cognitive rehabilitation in Ugandan pediatric cerebral malaria survivors. J Dev Behav Pediatr. 2009 Aug;30(4):310-8. doi: 10.1097/DBP.0b013e3181b0f01b. PMID 19668094
- [Background] John CC, Bangirana P, Byarugaba J, Opoka RO, Idro R, Jurek AM, Wu B, Boivin MJ. Cerebral malaria in children is associated with long-term cognitive impairment. Pediatrics. 2008 Jul;122(1):e92-9. doi: 10.1542/peds.2007-3709. Epub 2008 Jun 9. PMID 18541616
- [Background] Boivin MJ, Nakasujja N, Sikorskii A, Opoka RO, Giordani B. A Randomized Controlled Trial to Evaluate if Computerized Cognitive Rehabilitation Improves Neurocognition in Ugandan Children with HIV. AIDS Res Hum Retroviruses. 2016 Aug;32(8):743-55. doi: 10.1089/AID.2016.0026. Epub 2016 May 2. PMID 27045714
- [Background] Boivin MJ, Kakooza AM, Warf BC, Davidson LL, Grigorenko EL. Reducing neurodevelopmental disorders and disability through research and interventions. Nature. 2015 Nov 19;527(7578):S155-60. doi: 10.1038/nature16029. PMID 26580321
- [Derived] Boivin MJ, Sikorskii A, Nakasujja N, Ruisenor-Escudero H, Familiar-Lopez I, Opoka RO, Giordani B. Evaluating Immunopathogenic Biomarkers During Severe Malaria Illness as Modifiers of the Neuropsychologic Benefits of Computer Cognitive Games Rehabilitation in Ugandan Children. Pediatr Infect Dis J. 2019 Aug;38(8):840-848. doi: 10.1097/INF.0000000000002367. PMID 31232898
- See also: Webpage of the Makerere University/Michigan State University research collaboration — http://globalhealthuganda.org